CLINICAL TRIAL: NCT03956849
Title: Talking With Children About Weight and Lifestyle - Dutch Title: In Gesprek Over Gewicht en Leefstijl Met Kinderen
Brief Title: Talking With Children About Weight and Lifestyle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0931
Record Dates: First submitted 2019-05-01; First posted 2019-05-21 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Overweight and Obesity
Keywords: overweight; obesity; pediatric obesity
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Professionals working with children: The studypopulation for this mixed-methods study is consisting of healthcareprofessionals working with children (with overweight or obesity), such as pediatric residents, paediatricians and youth health care professionals. Also other professionals working with children, not working in the field of healthcare, such as teachers, can be included in the study population.
  Interventions: Other: Training COACH Conversationstarter

INTERVENTIONS:
Other: Training COACH Conversationstarter — After elaborating perceived barriers and facilitators via surveys and semi-structured focusgroups, a short training with the COACH Conversationstarter will be provided to a part of the participants. The COACH Conversationstarter will be provided to the participants attending the training, which they can use in the next couple of months. After a period of time all participants will be provided with a second questionnaire, and results of the group that received the COACH Conversationstarter will be compared with the group that didn't receive the COACH Conversationstarter. (A part of) the participants that used the COACH Conversationstarter will be interviewed about their experiences.
  However, the study will have an observational design, since the decision if a professional is attending the training is not based on the investigator / protocol, but depending on the professional, for example logistic reasons. This is part of routine education.

SUMMARY:
Obesity among children is a major problem. Therefore, it is important to start promoting a healthy lifestyle in an early stage. However, professionals find it difficult to start a conversation about overweight and lifestyle. Within Centre for Overweight Adolescent and Children's Healthcare (COACH) at the Maastricht University Medical Centre (MUMC+) a tool was developed, based on motivational interviewing, to help professionals engage in conversation with the children about weight and lifestyle.

The aim of this study is to identify barriers and facilitators perceived by professionals, working with children, to start a conversation with a child with overweight or obesity about weight and lifestyle. In addition, this study researches the effects of the developed COACH Conversationstarter, a tool that can help healthcare professionals to start a conversation with children about overweight and lifestyle and to gain more insight in the views, thoughts and beliefs of the child and its family.

DETAILED DESCRIPTION:
Overweight and obesity among children are major problems, not only in The Netherlands, but globally. Childhood obesity is associated with an increased risk for the development of different disease, like cardiovascular disease and sleep disorders, but it can also affect quality of life.

It's important to start promoting a healthy lifestyle among children and their parents in an early stage. The use of effective communication and respect to the language used is very important. However, international studies have shown that professionals experience barriers in starting a conversation about overweight and lifestyle. Examples of barriers may be fear of harm to the child, fear of parents' reactions and parents unmotivated to change. Knowledge regarding possible barriers and facilitators experienced specifically by Dutch healthcare professionals in talking about overweight is scarce.

National guidelines and the development of different visual tools (such as posters with pictures of healthy portion sizes and sugar amounts in beverages) are provided as facilitators in (visually) addressing lifestyle improvement by healthcare providers. However, they mainly focus on giving advice about creating a healthy lifestyle, rather than engaging in a conversation with children and parents about the current weight and lifestyle and exploring their views. In other words: these tools are developed to directly address the measures to be taken to change lifestyle, rather than discussing the status quo and exploring the underlying motivation. Within Centre for Overweight Adolescent and Children's Healthcare (COACH) at the Maastricht University Medical Centre (MUMC+) a tool was developed, based on motivational interviewing, to help professionals engage in conversation with children with overweight or obesity about weight and lifestyle.

The aim of this study is to identify barriers and facilitators perceived by healthcare professionals to start a conversation with a child about weight and lifestyle. In addition, this study researches the effects of the developed COACH Conversationstarter, a tool that can help healthcare professionals to start a conversation with children about overweight and lifestyle and to gain more insight in the views, thoughts and beliefs of the child and its family.

ELIGIBILITY:
Inclusion Criteria:

* Legally capable participants
* Professionals working with children
* Working with children between 8 - 17 years.
* To be willing to test the COACH Conversationstarter.

Exclusion Criteria:

* Professionals only working with children <8 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professionals working with children The studypopulation for this mixed-methods study is consisting of healthcareprofessionals working with children (with overweight or obesity), such as pediatric residents, paediatricians and youth health care professionals. Also other professionals working with children, not working in the field of healthcare, such as teachers can be included in the study population.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Barriers | January 2021
  Barriers perceived by the professionals to start a conversation about weight and lifestyle with children with overweight or obesity. Within the questionnaire a first selection of barriers will be made, which will be further in-depth explored in focusgroupinterviews.
Facilitators | January 2021
  Factors perceived as facilitator by the professionals to start a conversation about weight and lifestyle with children with overweight or obesity. Within the questionnaire a first selection of facilitators will be made, which will be further in-depth explored in focusgroupinterviews.
Experiences with the COACH Conversationstarter | January 2021
  Experiences with the COACH Conversationstarter, regarding design, usabilty and content. Within the questionnaire a first selection of experiences will be made, which will be further in-depth explored in semi-structured interviews.

SECONDARY OUTCOMES:
Level of participation | January 2021
  Percentage of time that each person (professional, parent(s) or child) is involved in a lifestyle-related conversation. Professionals can indicate the different percentages within the questionnaires.
Conversation skills | January 2021
  Confidence and thoughts about the own conversation skills of the professionals, for example regarding motivational interviewing. Measured within the questionnaire on a Likert-scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Vreugdenhil, Dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided